CLINICAL TRIAL: NCT01888133
Title: Adopting a Physically Active Lifestyle Through Organized Walk Events Among Joslin Clinic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, William Hsu, Director, Asian Clinic at Joslin Diabetes Center, Joslin Diabetes Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CHS 2012-12
Record Dates: First submitted 2013-04-02; First posted 2013-06-27 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Walk First (Experimental): Participants attend a weekly walking group session from weeks 1-6 and are not required to attend from weeks 7-12.
  Interventions: Behavioral: Group Walk; Behavioral: Individual Walk
- Individual Walk First (Experimental): Participants are not required to attend a weekly group walking sessions from weeks 1-6 and attend a weekly walking group session from weeks 7-12.
  Interventions: Behavioral: Group Walk; Behavioral: Individual Walk

INTERVENTIONS:
Behavioral: Group Walk — weekly walking club session on Saturday mornings at Boston Common, lasting 30 min - 1 hour and engage in daily physical activity (aiming for 10,000 steps/day or increase number of steps by 500 every 2 weeks)
Behavioral: Individual Walk — engage in daily physical activity (aiming for 10,000 steps/day or increase number of steps by 500 every 2 weeks)

SUMMARY:
Can participation in group physical activity, such as a community-based organized group walk, help adult diabetes patients develop a physically active lifestyle? Can such engagement ultimately lead to an improvement in hemoglobin A1c? To address this question, the investigators have designed this pilot study with the aim to investigate the effect of community-based group walks among Joslin adults with diabetes on the development of a physically active lifestyle and glycemic level. The investigators hypothesize that participation in group walking events helps Joslin adults with diabetes engage in physical activity and improves glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Joslin Clinic patients
* 18 years or older
* A1C between 7.5% - 12.0%
* Received physician clearance indicating safe to participate in the walk club events
* Reside within Boston and Greater Boston Area
* Ability to communicate in English and/or Chinese
* Agree to participate in the intervention walk club for 6 consecutive weeks

Exclusion Criteria:

* Pregnant or breast feeding
* Unstable angina or myocardial infarction within 1 month prior to screening
* Unstable gait, severe neuropathy, or deformed foot.
* Enrolled in another investigational study within 1 month prior to screening for this study
* On medications such as prednisone that will affect blood glucose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in steps/day | Baseline, Week 3, Week 6, Week 9, Week 12

SECONDARY OUTCOMES:
Change in BMI | Baseline, Week 3, Week 6, Week 9, Week 12
Change in Blood Pressure | Baseline, Week 3, Week 6, Week 9, Week 12
Change in Waist Circumference | Baseline, Week 3, Week 6, Week 9, Week 12
Hip Circumference | Baseline, Week 3, Week 6, Week 9, Week 12
Change in Physical Activity Pattern | Baseline, Week 6, Week 12
Change in Food Consumption | Baseline, Week 6, Week 12
Change in Fructosamine | Baseline, Week 6, Week 12
Change in Pulse | Baseline, Week 3, Week 6, Week 9, Week 12
Change in Height | Baseline, Week 3, Week 6, Week 9, Week 12
Change in Weight | Baseline, Week 3, Week 6, Week 9, Week 12
Change in A1c | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: William Hsu, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Tudor-Locke C, Bell RC, Myers AM, Harris SB, Ecclestone NA, Lauzon N, Rodger NW. Controlled outcome evaluation of the First Step Program: a daily physical activity intervention for individuals with type II diabetes. Int J Obes Relat Metab Disord. 2004 Jan;28(1):113-9. doi: 10.1038/sj.ijo.0802485. PMID 14569279
- [Background] Ford ES, Herman WH. Leisure-time physical activity patterns in the U.S. diabetic population. Findings from the 1990 National Health Interview Survey--Health Promotion and Disease Prevention Supplement. Diabetes Care. 1995 Jan;18(1):27-33. doi: 10.2337/diacare.18.1.27. PMID 7698044
- [Background] Hays LM, Clark DO. Correlates of physical activity in a sample of older adults with type 2 diabetes. Diabetes Care. 1999 May;22(5):706-12. doi: 10.2337/diacare.22.5.706. PMID 10332670
- [Background] Tudor-Locke CE, Bell RC, Meyers AM. Revisiting the role of physical activity and exercise in the treatment of type 2 diabetes. Can J Appl Physiol. 2000 Dec;25(6):466-92. doi: 10.1139/h00-031. PMID 11098158
- [Background] Manson JE, Hu FB, Rich-Edwards JW, Colditz GA, Stampfer MJ, Willett WC, Speizer FE, Hennekens CH. A prospective study of walking as compared with vigorous exercise in the prevention of coronary heart disease in women. N Engl J Med. 1999 Aug 26;341(9):650-8. doi: 10.1056/NEJM199908263410904. PMID 10460816
- [Background] Kang M, Marshall SJ, Barreira TV, Lee JO. Effect of pedometer-based physical activity interventions: a meta-analysis. Res Q Exerc Sport. 2009 Sep;80(3):648-55. doi: 10.1080/02701367.2009.10599604. No abstract available. PMID 19791652
- [Background] Merom D, Rissel C, Phongsavan P, Smith BJ, Van Kemenade C, Brown WJ, Bauman AE. Promoting walking with pedometers in the community: the step-by-step trial. Am J Prev Med. 2007 Apr;32(4):290-7. doi: 10.1016/j.amepre.2006.12.007. Epub 2007 Feb 15. PMID 17303369
- [Background] Kahn EB, Ramsey LT, Brownson RC, Heath GW, Howze EH, Powell KE, Stone EJ, Rajab MW, Corso P. The effectiveness of interventions to increase physical activity. A systematic review. Am J Prev Med. 2002 May;22(4 Suppl):73-107. doi: 10.1016/s0749-3797(02)00434-8. PMID 11985936
- [Background] American Diabetes Association. Executive summary: Standards of medical care in diabetes--2012. Diabetes Care. 2012 Jan;35 Suppl 1(Suppl 1):S4-S10. doi: 10.2337/dc12-s004. No abstract available. PMID 22187471
- [Background] Januszewski AS, Karschimkus C, Davis KE, O'Neal D, Ward G, Jenkins AJ. Plasma 1,5 anhydroglucitol levels, a measure of short-term glycaemia: assay assessment and lower levels in diabetic vs. non-diabetic subjects. Diabetes Res Clin Pract. 2012 Jan;95(1):e17-9. doi: 10.1016/j.diabres.2011.09.032. Epub 2011 Oct 22. PMID 22024285
- [Background] Barrett-Connor E. Nutrition epidemiology: how do we know what they ate? Am J Clin Nutr. 1991 Jul;54(1 Suppl):182S-187S. doi: 10.1093/ajcn/54.1.182S. PMID 2053559
- [Background] Lowe B, Kroenke K, Grafe K. Detecting and monitoring depression with a two-item questionnaire (PHQ-2). J Psychosom Res. 2005 Feb;58(2):163-71. doi: 10.1016/j.jpsychores.2004.09.006. PMID 15820844
- [Background] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035